CLINICAL TRIAL: NCT04062396
Title: Randomized Comparison Between Oxygenator Systems for the Reduction of Post-operative Delirium in Older Patients Undergoing Cardiac Surgery
Brief Title: Comparison of Remowell 2 and Inspire on Delirium and Cognitive Dysfunction
Acronym: CRIDD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maria Cecilia Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MCH2019-01
Record Dates: First submitted 2019-08-19; First posted 2019-08-20 (Actual); Last update posted 2024-02-20 (Actual); Status verified 2024-01

CONDITIONS: Cardiac Surgery; Cardiopulmonary Bypass

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Eurosets REMOWELL 2 oxygenator (Active Comparator)
  Interventions: Device: Eurosets REMOWELL 2 oxygenator
- LivaNova INSPIRE oxygenator (Active Comparator)
  Interventions: Device: LivaNova INSPIRE oxygenator

INTERVENTIONS:
Device: Eurosets REMOWELL 2 oxygenator — The main characteristic of REMOWELL 2 oxygenator is the presence of a filtration system for extracavitary inlet. Multilayer cascade filtration and supernatant separator leads to lipid-leukocytes depletion
  Arms: Eurosets REMOWELL 2 oxygenator
Device: LivaNova INSPIRE oxygenator — INSPIRE oxygenator has no filtration system for extracavitary inlet
  Arms: LivaNova INSPIRE oxygenator

SUMMARY:
Age is no longer an absolute contraindication to cardiac surgery therefore there is often need for combined interventions (double valve repair/replacement, or coronary artery bypass graft and valve repair/replacement) with relative prolongation of cardiopulmonary bypass time. Prolonged cardiopulmonary bypass use causes an increase in the inflammatory response, and on the other a need for blood reinfusion and therefore lipid microemboli from the operative field. The clinical consequences for patients are post-operative delirium and post-operative cognitive impairment.

These two neurological complications involve up to 45% of elderly patients undergoing cardiac surgery and have a significant impact on quality of life, hospitalization and mortality in the short and long term. The Remowell 2 oxygenator system has demonstrated in preliminary studies that, compared to the gold standard Inspire oxygenator, it can guarantee a significant reduction of hemodilution, inflammatory systemic response and embolization of lipid microemboli and leukocytes. In light of these considerations, it is possible to formulate the hypothesis that the use of the Remowell 2 device can contribute to significantly reducing the onset of post-operative delirium and cognitive impairment. The present study is designed to validate this hypothesis in a randomized controlled scenario.

ELIGIBILITY:
Inclusion Criteria:

1. Signature of informed consent for participation in the study
2. Age ≥65 years
3. Patients undergoing cardiac surgery of:

   1. coronary artery bypass graft and concomitant valve replacement/repair OR
   2. double valve replacement/repair

Exclusion Criteria:

1. Any documented history of cognitive impairment estimated as a mini mental state examination < 24 points
2. Patients who need blood prime in the cardiopulmonary bypass circuit
3. Chronic coagulopathies ( international normalized ratio > 2 in patients without anticoagulant treatment)
4. End stage renal disease on dialysis treatment
5. Previous cerebrovascular accident
6. Active cancer or immunological diseases
7. Liver cirrhosis (platelets <100.000/uL)
8. Decompensated diabetes
9. Severe preoperative anemia (hemoglobin <8 g/dl).

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 154 (Actual)
Dates: Start 2019-09-26 (Actual); Primary Completion 2023-01-23 (Actual); Study Completion 2023-01-23 (Actual)

PRIMARY OUTCOMES:
post-operative delirium | 6 days
  In-hospital incidence of post-operative delirium assessed by Confusion Assessment Method (CAM) diagnostic algorithm

CONTACTS AND LOCATIONS:
Overall Officials: Lorenzo Mantovani, MD, Principal Investigator — Maria Cecilia Hospital
Locations (1):
- Maria Cecilia Hospital, Cotignola, Ravenna, Italy

IPD SHARING:
Plan to Share IPD: Undecided